CLINICAL TRIAL: NCT00821938
Title: CRT in Patients With Narrow QRS, Echodesynchronisation and LV dp/Dt-Response With Pressure Wire
Brief Title: Cardiac Resynchronization Therapy (CRT)-Narrow-dp/Dt-Study
Acronym: CRT-Narrow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEN_G_CA_10
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2016-11

CONDITIONS: Heart Failure
Keywords: Narrow QRS; CRT
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRT-ICD (Active Comparator)
  Interventions: Procedure: LV dp/dt pressure measurement
- DDD-ICD (Placebo Comparator)
  Interventions: Procedure: LV dp/dt pressure measurement

INTERVENTIONS:
Procedure: LV dp/dt pressure measurement — Assessment of response to bi-ventricular pacing. Responder-arm, will be permanently paced bi-ventricularly
  Arms: CRT-ICD
Procedure: LV dp/dt pressure measurement — Assessment of response to bi-ventricular pacing. Non-esponder-arm, will be treated with standard ICD-treatment
  Arms: DDD-ICD

SUMMARY:
Goal is to examine the efficy of Cardiac Resynchronization Therapy in heart failure patients with narrow QRS complex and optimized medical treatment but echocardiographic desynchronization detection as well as the positve increase of the intraoperative pressureincreasespeed in reverse remodelling and a secondary improvement of functional parameters

ELIGIBILITY:
Inclusion Criteria:

* EF < 35%
* CHD or dilate cardiomyopathy
* sinus rhythm
* NYHA III (or IV but stable recompenstated)
* QRS < 120 ms 2-3 of the following:
* LV-fillingtime < 40% of the cyclelength
* TDI septal-lateral (LV basal) > 60ms
* 2D-Strain-Score > 9 points

Exclusion Criteria:

* tricuspid or artificial valve
* AV block II or III or PQ time > 250ms
* revasculisation or condition after cardiac surgery < 3 months
* myocardial infarction or bypass OP < 3 months
* hytertrphic obstructive cardiomyopathy, constrictive pericarditis
* intravenous catecholamines because of HF
* manifeste hyperthyreoses
* kidney failure (creatine >2,5 mg/dl)
* no written informed consent
* no compliance
* participation in another study
* life expectancy < 1 year
* patients < 18 years
* pragnancy or no safe contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2012-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Indexed left ventricular volume | 12 months

SECONDARY OUTCOMES:
NYHA-class, 6 minute hallwalk, QOL, BNP-level, echo-criteria | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Guido Luedorff, MD, Principal Investigator — Schuechtermann-Kliniken
Locations (1):
- Schuechtermann-Kliniken, Bad Rothenfelde, Germany